CLINICAL TRIAL: NCT03725423
Title: Apatinib Mesylate Was Used in the Treament of Patients With Advanced Lung Squamous Cell Carcinoma of the Third Line and Above
Brief Title: Apatinib for Advanced Lung Squmamous Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Feng Chunguang, Chief Physician, Xuzhou Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XuzhouCH
Record Dates: First submitted 2018-10-25; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Lung Squamous Cell Carcinoma
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Oral administration of 250mg of apatinib daily, with or without chemotherapy
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 250mg, qd once a day, take it half an hour after meal (the time for taking the medicine should be the same as possible), and take it with warm water. 28 days is a drug delivery cycle.

SUMMARY:
In order to search for effective and low toxicity anti-tumor angiogenesis drugs, jiangsu hengrui pharmaceutical co., ltd. developed the high-efficiency VEGFR2 tyrosine kinase inhibitor apatinib. This drug is mainly used to treat malignant tumors by inhibiting VEGFR2 to play an anti-angiogenic role. Both in vivo and in vitro experiments have shown that apatinib has good tumor growth inhibition activity for lung cancer. This study aims to further confirm the effectiveness and safety of apatinib third-line treatment for patients with advanced lung squamous cell carcinoma.

DETAILED DESCRIPTION:
Apatinib, 250mg, once a day (qd), take it half an hour after meal (the time for taking the medicine should be the same as possible), and take it with warm water. 28 days is a drug delivery cycle.According to the patient's condition, a single drug was selected for 6 cycles of chemotherapy in gemcitabine, yew and ruibin, changchun. After the chemotherapy, the single drug apatinib was maintained.Adverse reactions should be closely monitored during the use of apatinib and adjusted as needed to enable patients to tolerate treatment. The adverse reactions caused by apatinib can be treated by symptomatic treatment, drug withdrawal and dose adjustment. In clinical studies, dose adjustment usually occurs in the second and third cycles (28 days is one cycle). In case of 3/4 grade adverse reactions, the drug can be suspended until the toxic and side effects are completely recovered. Exit the study if 3/4 level of adverse reactions occur again after resumption of medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age: more than 18 years old;
2. The pathology diagnosed late (Ⅲ B, Ⅳ) lung squamous cell carcinoma, with measurable lesion (tumor lesions on CT scan length to diameter 10 mm, or lymph node lesions on CT scans short diameter 15 mm or higher, scanning is not more than 5 mm, with a thick layer of measurable lesions not received radiotherapy, refrigeration, etc).
3. Patients who have been treated with Eastern Cooperative Oncology Group for recurrence or failure of at least two-line standard treatment can be enrolled; Definition of "treatment failure" :(1) clear imaging or clinical evidence of disease progression during or after the last treatment; (2) could not be intolerance events out of the standard treatment by CTCAE 4.0 standard, the intolerance of adverse events mean acuity level Ⅳ hematology toxicity or acuity levels Ⅲ non hematologic toxicity or acuity Ⅱ heart, liver, kidney and other major organs damage.
4. Eastern Cooperative Oncology Group score: 0-2;
5. The predicted survival time is greater than or equal to 3 months;
6. The damage caused by other treatments has been recovered (nci-ctcae version 4.0 grade is no more than 1), and the interval between receiving nitro-urea or mitomycin is no more than 6 weeks; Other cytotoxic drugs, Avastin, radiotherapy or surgery were performed for 4 weeks or longer. Eastern Cooperative Oncology Group TKI molecular targeted drugs were more than 2 weeks old;
7. Normal function of the main organs means that the following criteria are met:

(1) blood routine examination standards shall be met (no blood transfusions and blood products within 14 days, no g-csf and other hematopoietic stimulant correction is performed) :hb≥90 g / L;b . anc≥1.5×109 / L;c . plt≥80×109 / L; (2)biochemical test shall meet the following standards:

1. total bilirubin<1.5upper limit of normal;
2. ALT and AST<2.5upper limit of normal, and < 5upper limit of normal for patients with liver metastasis;
3. Serum Cr is no more than 1.25upper limit of normal or Endogenous creatinine clearance rate > 45 ml/min (Cockcroft-Gault formula); 8. Women of childbearing age must have had access to reliable contraception or to a pregnancy test (serum or urine) within 7 days of enrollment with negative results and be willing to use an appropriate method of contraception eight weeks after the trial period and the last time the trial drug was administered. For men, consent should be given to use an appropriate method of contraception or surgical sterilization eight weeks after the trial period and the last administration of the drug; 9. The subjects voluntarily joined the study and signed the informed consent, with good compliance and followed up.

Exclusion Criteria:

1. Cancer meningitis, spinal cord compression, or screening imaging CT or MRI found brain or pial meninges disease (21 days before the treatment and stable symptoms of brain metastases can be admitted to the group, but only through brain MRI, CT or venography were confirmed as anencephalic hemorrhage symptoms.
2. Patients with symptomatic central nervous system metastasis.
3. Imaging (CT or MRI) showed that the tumor focus was no more than 5 mm from the large blood vessels, or there was a central tumor invading the local large blood vessels.
4. Uncontrolled hypertension (systolic blood pressure of 140mmhg or diastolic pressure of 90mmhg, despite the best drug treatment);
5. Suffering from myocardial ischemia and myocardial infarction Ⅱ class above, poor control of arrhythmia (including QTc interphase male 450, female 470 ms or ms or higher);
6. According to NYHA standard Ⅲ ~ Ⅳ cardiac insufficiency, or heart colour to exceed revealed left ventricular ejection fraction (LVEF) < 50%;
7. Abnormal coagulation function (INR >1.5 or prothrombin time (PT) > upper limit of normal+4 seconds or APTT >1.5upper limit of normal), with bleeding tendency or being treated with thrombolysis or anticoagulation;
8. Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs; Note: under the premise that the internationally standardized ratio (INR) of prothrombin time is no more than 1.5, low doses of heparin (60 thousand to 12 thousand U per day for adults) or low doses of aspirin (no more than 100 mg per day) are allowed for preventive purposes.
9. Significant hemoptysis, or hemoptysis, of half a teaspoon (2.5ml) or more per day within 2 months before enrollment;
10. Bleeding symptoms with significant clinical significance or with definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood at baseline ++ and above, or with vasculitis, etc. appear within 3 months before enrollment;
11. Arteriovenous thrombosis events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. occurred within 12 months before enrollment;
12. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., haemophiliacs, clotting disorders, thrombocytopenia, hypersplenism, etc.);
13. Long term untreated wounds or fractures;
14. Received major surgery or developed severe traumatic injury, fracture or ulcer within 4 weeks before enrollment;
15. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
16. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before enrollment;
17. The routine urine test suggested that the urine protein was greater than or equal to ++, or the 24-hour urine protein was greater than or equal to 1.0g.
18. Patients with active viral hepatitis b or c;
19. Active infections that require antimicrobial treatment (e.g. antimicrobial, antiviral, antifungal);
20. Persons who have a history of psychotropic drug abuse and are unable to quit or have mental disorders;
21. Participated in other clinical trials of anti-tumor drugs within 4 weeks before enrollment;
22. Before entering into the group, I used the inhibitor of the Vascular epidermal growth factor (except bevacizumab);
23. Previous or concurrent incurable malignancies, with the exception of cured basal cell carcinoma of the skin, in situ carcinoma of the cervix and superficial bladder cancer;
24. Those who had been treated with strong CYP3A4 inhibitor within 7 days before enrollment, or who had been treated with strong CYP3A4 inducer within 12 days before participating in the study;
25. Pregnant or lactating women; A person who is unable or unwilling to take effective contraceptive measures;
26. The investigator identifies other conditions that may affect the conduct of clinical studies and the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Respond Evaluation Criteria in Solid Tumors | Through study completion,an average of 1 year
  Complete Response, partial response

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wang, Master, Principal Investigator — Xuzhou central hospaital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davies H, Hunter C, Smith R, Stephens P, Greenman C, Bignell G, Teague J, Butler A, Edkins S, Stevens C, Parker A, O'Meara S, Avis T, Barthorpe S, Brackenbury L, Buck G, Clements J, Cole J, Dicks E, Edwards K, Forbes S, Gorton M, Gray K, Halliday K, Harrison R, Hills K, Hinton J, Jones D, Kosmidou V, Laman R, Lugg R, Menzies A, Perry J, Petty R, Raine K, Shepherd R, Small A, Solomon H, Stephens Y, Tofts C, Varian J, Webb A, West S, Widaa S, Yates A, Brasseur F, Cooper CS, Flanagan AM, Green A, Knowles M, Leung SY, Looijenga LH, Malkowicz B, Pierotti MA, Teh BT, Yuen ST, Lakhani SR, Easton DF, Weber BL, Goldstraw P, Nicholson AG, Wooster R, Stratton MR, Futreal PA. Somatic mutations of the protein kinase gene family in human lung cancer. Cancer Res. 2005 Sep 1;65(17):7591-5. doi: 10.1158/0008-5472.CAN-05-1855. PMID 16140923